CLINICAL TRIAL: NCT04810442
Title: Investigation of Neural Mechanisms Associated With Sleep-Dependent Enhancement of Motor Learning After Brain Injury
Brief Title: Investigating How Sleep After Training Can Affect the Learning of a Motor Skill in Individuals With Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R-1061-19
Record Dates: First submitted 2019-12-05; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Traumatic Brain Injury
Keywords: functional MRI; Motor Learning; Nap; Sleep Benefits; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nap Group (Experimental): This group will be involved with taking a nap in between the two scanning procedures.
  Interventions: Other: Nap
- No-Nap Group (No Intervention): This group will not be taking a nap in between the two scanning procedures, and instead will be silently watching a film for the 45 minute period.

INTERVENTIONS:
Other: Nap — 45-minute nap between scanning procedures
  Arms: Nap Group

SUMMARY:
Studies have shown that a period of sleep, even in the form of a daytime nap, after a period of training on a motor learning task can boost subsequent performance beyond that observed after an equal amount of time spent awake and resting. This leap in performance has been referred to as "off-line" motor learning because it occurs during a period of sleep in the absence of additional practice. Motor learning is an integral part of the physical and occupational therapy that patients receive after traumatic brain injury (TBI) in which various activities of daily living may need to be relearned. Targeted motor skills may include dressing (learning how to zip up a jacket or button a shirt), using a fork and knife to eat, or using technology (tapping touch screen on a cell phone or typing on a computer). Yet the potential of sleep in the form of a strategic nap as a therapeutic tool to maximize motor learning in rehabilitation therapies has not been fully realized. In addition, a growing body of research among healthy individuals has shown evidence of changes in the brain associated with enhanced performance among those who slept following training compared with those who spent the same amount of time awake. The neural mechanisms of "off-line" motor learning have not been studied among individuals with TBI. Using functional neuroimaging and measurement of brain waves, the current study will examine the mechanisms underlying this sleep-related enhancement of motor learning among individuals with TBI and determine how brain physiology may influence the magnitude of the effect. By understanding how this treatment works and identifying the factors that modulate its effectiveness we can identify which individuals will be most likely to benefit from a nap after training to improve motor learning after TBI. This can provide a more person-centered approach to treatment delivery that can maximize the effectiveness of a simple but potent behavioral intervention.

DETAILED DESCRIPTION:
Procedural memory is vitally important to the efficacy of rehabilitation following Traumatic Brain Injury (TBI). Specifically, during rehabilitation, persons with TBI must re-learn many motor skills associated with activities of daily living to improve functional outcomes. Emerging research on neuroplasticity after brain damage is beginning to increase our understanding of motor learning principles and how they interact with the training that takes place in neurorehabilitation.

There is a strong body of evidence showing the importance of sleep in procedural learning among healthy individuals. Within this body of research on sleep and procedural learning, there is substantial evidence demonstrating sleep-dependent neuroplasticity. Participants trained on a motor learning task show improvements over the training period, as expected. However, when re-tested after a period of sleep, performance is significantly better than when retested after an equivalent period of time awake. The actual enhancement of a learned motor skill in the absence of additional practice trials suggests that one can decrease the time necessary for learning a motor skill by incorporating a daytime nap after a period of training. The implications of these findings can be ground-breaking when applied to brain injury rehabilitation where motor learning may be a major focus of physical and occupational therapies. There is evidence of a positive impact of sleep on procedural memory and rehabilitation progress among older individuals after stroke, and the investigators have pilot data showing a substantial positive effect of a post-training nap on motor learning in an acquired brain injury sample. However, the neural mechanisms involved in this process after traumatic brain injury are less understood.

Among healthy individuals, there are numerous studies examining neural biomarkers that can quantify the effect of sleep on motor learning. Studies have reported that changes in sleep physiology and neural activation after training correlate with the degree of improvement at post-intervention testing. Studies showed that, after a nap of 60-90 minutes, speed of performance was enhanced, and the degree of enhancement was associated with the duration of stage 2 non-rapid eye movement (NREM) sleep. This relationship with stage 2 NREM sleep has also been shown after a 20-minute nap. In addition, changes in neural activation in the striatum have been found to be more pronounced when individuals slept after training than when they remained awake. In another study in which a night of sleep occurred between training and retest, changes in striatal activity were correlated with performance gains on the motor learning task. This study also showed evidence of EEG changes during sleep after the training period in the amount of sleep-spindle activity, a waveform associated with stage 2 NREM sleep.

While our preliminary findings show evidence of off-line motor learning after a nap among individuals with acquired brain injury, research into the mechanisms of action driving this response among individuals with TBI is lacking. A better understanding of neurophysiology and its influence on the magnitude of the effect is a crucial step in determining which individuals would be likely to benefit from this behavioral intervention.

Specific Aim 1-Behavioral Intervention: In a sample of individuals with TBI living in the community, demonstrate greater improvement on a motor sequence learning task after a daytime nap compared with an equivalent time spent awake and resting. This aim will also explore the individual differences in terms of demographics and injury characteristics contributing to the magnitude of the effect.

Hypothesis 1. Individuals exposed to a nap after a period of training on the motor sequence learning task will demonstrate greater improvement in speed and accuracy from the end of training to the post-nap retesting.

Research Question 1. How does the magnitude of the effect correlate with demographic factors and injury characteristics? Specific Aim 2-Functional Neuroimaging: To examine the neural correlates of off-line motor learning among individuals with TBI who were given a nap after training on the motor sequence learning task using functional MRI compared with a control group who received an equivalent period of time awake.

Hypothesis 2. Individuals in the nap group will show more pronounced changes in activation within the striatum and motor cortex compared with those who remained awake and resting.

Specific Aim 3-Sleep Physiology: To examine aspects of stage 2 sleep associated with performance gains (duration of stage 2 and degree of spindle activity) occurring during the nap period after training.

Hypothesis 3a. Among participants in the nap group, there will be a significant positive correlation between the degree of improvement and the duration of stage 2 sleep.

Hypothesis 3b. Among participants in the nap group, there will be a significant positive correlation between the degree of improvement and density of sleep spindles.

ELIGIBILITY:
Inclusion Criteria:

* I am between the ages of 18-65
* I have a diagnosis of a moderate to severe Traumatic Brain Injury
* I am at least 1 year post-injury
* I am a habitual napper (I nap at least once per week) or I am able to fall asleep in a comfortable reclining chair in a dimly lit room
* I am right handed
* I can read and speak English fluently

Exclusion Criteria:

* I am pregnant
* I have had a prior stroke or neurological disease
* I have a history of significant psychiatric illness
* I am unable to demonstrate fine motor movements by touching each of my fingers to my thumb on the same hand
* I am taking dopaminergic medication.
* I have a significant alcohol or drug abuse history
* My vision is impaired - more than 20/60 in worst eye
* I have previous experience in playing a musical instrument
* I have been told by my doctor that it is unsafe for me to receive regular MRI
* I have non-titanium metal in my body or something in my body in which will keep me from being still in the MRI
* I have a movement disorder in which will keep me from being still in the MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Tapping Task Performance Gain | through study completion, an average of 2 years
  The number of correct tapping sequences across 30sec time intervals for the learning trials and post-intervention retest trials will be calculated for each participant. Tapping Task Performance Gain will be operationally defined as the mean of correct sequences within the final block of learning trials subtracted from the mean of correct sequences within the first block of retest trials. Analysis of Covariance will be performed with Tapping Task Performance Gain as the independent variable and treatment group (Nap vs. Rest) as the dependent variable. Covariates of age and learning capacity (calculated as the difference between the mean of correct sequences in the initial and final blocks of the learning trials) will be entered into the model.
Bold Signal Change | through study completion, an average of 2 years
  Beta weights associated with the Nap and Rest Groups.
Number of Sleep Spindles | through study completion, an average of 2 years
  The number of sleep spindles in the EEG output generated by the Sleep Profiler within the 45-minute nap will be counted. Pearson correlations will be used to examine the relationship between performance gains and the number of sleep spindles within the Nap group.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lequerica, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleim JA. Neural plasticity and neurorehabilitation: teaching the new brain old tricks. J Commun Disord. 2011 Sep-Oct;44(5):521-8. doi: 10.1016/j.jcomdis.2011.04.006. Epub 2011 Apr 30. PMID 21600589
- [Background] Krakauer JW. Motor learning: its relevance to stroke recovery and neurorehabilitation. Curr Opin Neurol. 2006 Feb;19(1):84-90. doi: 10.1097/01.wco.0000200544.29915.cc. PMID 16415682
- [Background] Nudo RJ. Neural bases of recovery after brain injury. J Commun Disord. 2011 Sep-Oct;44(5):515-20. doi: 10.1016/j.jcomdis.2011.04.004. Epub 2011 Apr 30. PMID 21600588
- [Background] Smith C, MacNeill C. Impaired motor memory for a pursuit rotor task following Stage 2 sleep loss in college students. J Sleep Res. 1994 Dec;3(4):206-213. doi: 10.1111/j.1365-2869.1994.tb00133.x. PMID 10607127
- [Background] Walker MP, Brakefield T, Morgan A, Hobson JA, Stickgold R. Practice with sleep makes perfect: sleep-dependent motor skill learning. Neuron. 2002 Jul 3;35(1):205-11. doi: 10.1016/s0896-6273(02)00746-8. PMID 12123620
- [Background] Walker MP, Stickgold R, Alsop D, Gaab N, Schlaug G. Sleep-dependent motor memory plasticity in the human brain. Neuroscience. 2005;133(4):911-7. doi: 10.1016/j.neuroscience.2005.04.007. PMID 15964485
- [Background] Walker MP. Sleep-dependent memory processing. Harv Rev Psychiatry. 2008;16(5):287-98. doi: 10.1080/10673220802432517. PMID 18803104
- [Background] Walker MP, Stickgold R. Sleep, memory, and plasticity. Annu Rev Psychol. 2006;57:139-66. doi: 10.1146/annurev.psych.56.091103.070307. PMID 16318592
- [Background] Milner CE, Fogel SM, Cote KA. Habitual napping moderates motor performance improvements following a short daytime nap. Biol Psychol. 2006 Aug;73(2):141-56. doi: 10.1016/j.biopsycho.2006.01.015. Epub 2006 Mar 15. PMID 16540232
- [Background] Korman M, Doyon J, Doljansky J, Carrier J, Dagan Y, Karni A. Daytime sleep condenses the time course of motor memory consolidation. Nat Neurosci. 2007 Sep;10(9):1206-13. doi: 10.1038/nn1959. Epub 2007 Aug 12. PMID 17694051
- [Background] Siengsukon CF, Boyd LA. Sleep enhances implicit motor skill learning in individuals poststroke. Top Stroke Rehabil. 2008 Jan-Feb;15(1):1-12. doi: 10.1310/tsr1501-1. PMID 18250068
- [Background] Nishida M, Walker MP. Daytime naps, motor memory consolidation and regionally specific sleep spindles. PLoS One. 2007 Apr 4;2(4):e341. doi: 10.1371/journal.pone.0000341. PMID 17406665
- [Background] Backhaus J, Junghanns K. Daytime naps improve procedural motor memory. Sleep Med. 2006 Sep;7(6):508-12. doi: 10.1016/j.sleep.2006.04.002. Epub 2006 Aug 23. PMID 16931152
- [Background] Debas K, Carrier J, Orban P, Barakat M, Lungu O, Vandewalle G, Hadj Tahar A, Bellec P, Karni A, Ungerleider LG, Benali H, Doyon J. Brain plasticity related to the consolidation of motor sequence learning and motor adaptation. Proc Natl Acad Sci U S A. 2010 Oct 12;107(41):17839-44. doi: 10.1073/pnas.1013176107. Epub 2010 Sep 27. PMID 20876115
- [Background] Fogel S, Albouy G, King BR, Lungu O, Vien C, Bore A, Pinsard B, Benali H, Carrier J, Doyon J. Reactivation or transformation? Motor memory consolidation associated with cerebral activation time-locked to sleep spindles. PLoS One. 2017 Apr 19;12(4):e0174755. doi: 10.1371/journal.pone.0174755. eCollection 2017. PMID 28422976